CLINICAL TRIAL: NCT02023632
Title: A Self-categorization Theory Approach to Fostering Physical Activity Adherence Among Older Adults: A Randomized Controlled Feasibility Trial.
Brief Title: GrOup-based Physical Activity for oLder Adults Trial
Acronym: GOAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H13-01593; DCO150GP (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-12-17; First posted 2013-12-30 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Motor Activity
Keywords: older adults; physical activity; self-categorization; group dynamics; self-identity
MeSH Terms: conditions — Motor Activity | interventions — methyl alpha-D-6-(12-(9-anthroyl)stearoyl)glucoside

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Similar-Age-Same-Gender (SASG) (Experimental): Participants in this trial arm will be of similar age (65+) and of the same gender (i.e., separate groups for male older adults and female older adults).
  Interventions: Behavioral: Similar-Age-Same-Gender (SASG)
- Similar-Age-Mixed-Gender (SAMG) (Active Comparator): This group will include participants of both genders who are similar aged (65+).
  Interventions: Behavioral: Similar-Age-Mixed-Gender (SAMG)
- Mixed-Age-Mixed-Gender (MASG) (Sham Comparator): This group is used as the 'standard' group based exercise course; including those of mixed age and mixed gender.
  Interventions: Behavioral: Mixed-Age-Mixed-Gender (MASG)

INTERVENTIONS:
Behavioral: Similar-Age-Same-Gender (SASG) — The core feature of the program is that it is exclusively for those of a similar age and same gender. Such an environment was reported to provide opportunities for social connectedness, as well as personal comfort. Secondly, exercise class instructors are volunteers- both providing 'similar-models' to enhance efficacy as well as reduce costs associated with instructors. Consistent with social identity and self-categorization perspectives, the program also makes use of a series of strategies to foster intra-group attraction and group identity. For many of the participants a major draw of the program is that it provides opportunities for the older adults to connect with one another after the classes have ended.
  Arms: Similar-Age-Same-Gender (SASG)
Behavioral: Similar-Age-Mixed-Gender (SAMG) — The SAMG physical activity condition will mirror the SASG group condition, but will be open to older adults from both genders. The same strategies to those used within the SASG condition will also be utilized (development of a unique program name, T-shirts, opportunities to socialize after the program), and will be offered three days per week (Mon, Wed, Fri, or Tues, Thurs, Sat). Older adults will also be recruited to be instructors for the group classes (= 65 years), with both males and females invited to occupy these instructional roles. (As with the SASG condition, training will take place between September and December 2013, through the respective YMCA centres. The YMCA will oversee the training of these volunteers through their Fitness Leader Training Program).
  Arms: Similar-Age-Mixed-Gender (SAMG)
Behavioral: Mixed-Age-Mixed-Gender (MASG) — The third condition utilized within the RCT is designed to reflect 'standard' group based exercises that one sees in typical physical activity centres. Specifically, these classes are not restricted to participants on the basis of age or gender, and as such older adults will be participating in groups comprised of people younger than themselves as well as those of both gender.
  Arms: Mixed-Age-Mixed-Gender (MASG)

SUMMARY:
Regular physical activity is associated with a diverse range of physical and mental health outcomes, with the effects being particularly pronounced among older adults. Despite these health benefits, involvement in physical activity has been found to decline over the course of adulthood with older adults in particular risk of inactivity. A growing body of evidence, however, suggests that group-based settings that are sensitive to both the age-composition and gender-composition of their constituent members may represent an opportune means of supporting the improved adoption and maintenance of older adults in physical activity programs. The overall purpose of this feasibility trial is to test the effectiveness of a group-based physical activity program for older adults that is sensitive to both age-congruent and gender-congruent contextual factors, in supporting their sustained involvement in physical activity.

DETAILED DESCRIPTION:
The results of prominent meta-analytic reviews suggest that when people exercise in groups they tend to sustain their involvement to a greater extent than when they exercise on their own. Despite the potential for groups to sustain long-term physical activity behaviours, there appears to be an important caveat that comes with exercising with others: if people perceive themselves to be similar to other members of a given group, in terms of salient underlying qualities, this corresponds positively with their attraction to, and level of involvement within, that group. If, however, people perceive themselves to be distinctly different from others within their social group, this is likely to undermine their attraction to, and involvement in that group. Recent research by Dr. Beauchamp and his team suggests that across the adult age spectrum people report a positive preference for exercising within groups that are comprised of others their own age, and when they participate in such classes they display higher levels of adherence to the group. In a similar regard, people report comparable positive preferences for same-gender rather than mixed-gender physical activity group settings. However, to date, research has yet to examine these effects using an experimental (RCT) design. This constitutes the purpose of this present trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 65 years of age or older (both males and females), be able to speak and read English, and not experience any contraindication which might prevent that person from participating in moderate-intensity physical activity. Participants will be required to complete PAR-Q+, and where necessary ePARmed-X.

Exclusion Criteria:

* The only exclusionary criteria is that participants must be 65 years of age or older (both males and females), be able to speak and read English, and not experience any contraindication which might prevent that person from participating in moderate-intensity physical activity.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 554 (Actual)
Dates: Start 2014-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Program adherence and re-enrollment | Month 3 (May 2014;2015) and Month 6 (August 2014;2015)
  Physical activity centre records (i.e., the YMCA) will be utilized to provide an objective measure of class attendance through "signing-in". With regard to the secondary research question concerning the extent to which participants choose to re-enroll after the initial 3-month program has ended, program enrollment records will again be used.

SECONDARY OUTCOMES:
Change in Cohesion | Weeks 2, 7, 12, 14, 19, 24
  Class cohesion will be assessed using the Physical Activity Group Environment Questionnaire (PAGEQ. The PAGEQ is a 21-item self-report questionnaire designed to assess four dimensions of cohesion within exercise classes; namely, attraction to the group's task (ATG-T), and social (ATG-S) activities, as well as perceptions of group integration around the group's task (GI-T), and social (GI-S) activities. The PAGEQ was developed (by Dr. Estabrooks, Co-I) specifically with older adults in mind taking part in physical activity classes such as those involved in this trial, with scores derived from this instrument demonstrating good reliability (α ≥ .72), factorial validity, and predictive utility.
Change in Affective and Instrumental Attitudes | Weeks 2, 7, 12, 14, 19, 24
  Affective attitudes towards physical activity will be assessed using the procedures outlined by Ajzen (2002). Specifically, a 7-point semantic differential scale will be used, with anchors including "Enjoyable-Unenjoyable", "Pleasant-Unpleasant", "Interesting-Boring". Previous research with older adults has found support for both the internal consistency and predictive utility of scores derived from this instrument.
Physical Health Screening Measure | Prior to the start of the program (February 2014 and December 2014/January 2015)
  For pre-screening all individuals will complete the Physical Activity Readiness Questionnaire for everyone (PAR-Q+). If participants respond 'NO' to all of the (seven) questions within the PAR-Q+ they are cleared for participation in physical activity. If participants have a positive response to the PAR-Q+ (e.g., due to a current medical condition), participants automatically proceed to a second series of questions subsumed within the ePARmed-X. As a result of completing the ePARmed-X, they will either be cleared for participation in physical activity OR will be directed to their physician to obtain clearance before they can participate in physical activity. If older adults have a medical contraindication (flagged through the PAR-Q+ and ePARmedX) and have NOT been cleared to participate in physical activity by their physician they are then ineligible to participate in the study.
Change in Self-efficacy | Weeks 2, 7, 12, 14, 19, 24
  During the program, in-class task self-efficacy will be measured through a validated and reliable measure (Poag-Ducharme & Brawley, 1993). Self-efficacy to overcome barriers to exercise (with an emphasis on self-regulation) will use Bray and colleagues (2001) validated and reliable measure; using 0-100% confidence. An example self-efficacy question is: how confident they may be in "Completing the warm-up and stretching component of each class."
Change in Stigma Consciousness | Weeks 2, 7, 12, 14, 19, 24
  To measure both gender and ethnicity stigma, we will use Pinel's (1999) measure for "stigma consciousness." Each item is on a 6-point Likert scale. An example item is "I never worry that I will be viewed as being stereotypically [fe]male."
Change in Flourishing | Weeks 2, 7, 12, 14, 19, 24
  Diener et al's(2009) well-being measure of the relationship of flourishing and positive and negative feelings will be distributed post-class at each of the times listed above. This measure is on a 7-point Likert scale from strongly disagree to strongly agree with items such as "I am engaged and interested in my daily activities" and "I am a good person and live a good life."
Change in Perceptual Similarity | Weeks 2, 14
  Using methods from Beauchamp et al (2012), participants will answer a series of questions regarding their perceived similarity via a 9-point Likert scale. Surface-level perceptions will be assessed through items related to age, physical condition, and physical appearance similarity, whereas deep-level perceptions will be assessed through items related to attitude, belief, and value similarity. Exemplar items from this assessment included, "In my exercise class, I believe members are similar to me in terms of age."
Change in commute time and commute mode | Weeks 2 and 14
  Two-item assessment of how participants commute to the YMCA location: 1. Typically, how long does it take for you to get to your physical activity class (i.e., commute time):________________ mins and 2) What mode of transport do you use to get to your physical activity class (car, bus, bike, train, walk, taxi):_____________________.
Change in Group-Interaction Variables | Weeks 7 and 19
  To measure the group-interaction variables of interest (i.e., communication, cooperation, and competition) additional items are embedded within the PAGEQ. Communication will be measured through 6 items that can be further divided into task communication (e.g., 'members of our group talk about how often they should do physical activity') and social communication (e.g., 'people of this group talk about things that are happening in our lives'). Cooperation will be measured through 3 items (e.g., 'we all cooperate to help this group's program run smoothly') as will competition (e.g., 'There is friendly competition within the members to stay as healthy as possible'). Internal consistencies for the group-interaction variables were all previously acceptable: task communication (α = .94), social communication (α = .65), cooperation (α = .91), and friendly competition (α = .81) (Harden, Mama, Lee, Estabrooks, Under Review).
Change in Physical Activity Outside of the YMCA | Week 12, 24
  Physical activity outside of program will be measured by an adapted 3-step procedure outlined by Wilcox et al. (1999), specific for older adults. Participants will report on various activities that they engaged in over the last two weeks as well as how many times and the duration associated with each. Participants will also answer whether they experienced (a) no, (b) small, (c) moderate, or (d) large increases in heart and breathing rates while participating.
Change in Functional Fitness Appraisal | Prior to the start of the program (February 2014, January 2015) and after the end of the program (August 2014, 2015)
  Functional fitness testing will be conducted based on a previously developed and validated functional fitness test for community-residing older adults (Rikli, R. E., & Jones, C. J. 1999). The assessment will include measures of upper and lower body strength and flexibility, aerobic endurance, dynamic balance, and Body Mass Index. These tests will be done at the participant's local YMCA by trained research assistants.

OTHER OUTCOMES:
Process Evaluation | After the end of the program (August 2014, 2015)
  The process evaluation procedures to be used in this study first involves identifying fidelity to the five key components of the intervention. Second, semi-structured interviews will be used that allow us to examine each of the subcomponents described in the first step. Interviews will be conducted with participants by trained research assistants, and although qualitative data analysis will be overseen by the principal investigator, the coding will be performed by research assistants (i.e., unconnected with the intervention activities).

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Beauchamp, PhD, Principal Investigator — University of British Columbia
Locations (3):
- Canada (3):
  - Surrey Family YMCA, Surrey, British Columbia
  - Langara YMCA, Vancouver, British Columbia
  - Robert Lee YMCA, Vancouver, British Columbia

REFERENCES:
- [Background] Dunlop WL, Beauchamp MR. Birds of a feather stay active together: a case study of an all-male older adult exercise program. J Aging Phys Act. 2013 Apr;21(2):222-32. doi: 10.1123/japa.21.2.222. Epub 2012 Aug 14. PMID 22899819
- [Background] Rikli RE, Jones CJ. Functional fitness normative scores for community-residing older adults, ages 60-94. Journal of aging and physical activity 7:162-181, 1999.
- [Background] Beauchamp M, Dunlop WL, Downey SM, Estabrooks PA. First impressions count: perceptions of surface-level and deep-level similarity within postnatal exercise classes and implications for program adherence. J Health Psychol. 2012 Jan;17(1):68-76. doi: 10.1177/1359105311408156. Epub 2011 Jun 6. PMID 21646291
- [Background] Dunlop WL, Beauchamp MR. The relationship between intra-group age similarity and exercise adherence. Am J Prev Med. 2012 Jan;42(1):53-5. doi: 10.1016/j.amepre.2011.08.018. PMID 22176846
- [Background] Beauchamp MR, Carron AV, McCutcheon S, Harper O. Older adults' preferences for exercising alone versus in groups: considering contextual congruence. Ann Behav Med. 2007 Apr;33(2):200-6. doi: 10.1007/BF02879901. PMID 17447872
- [Background] Dunlop WL, Beauchamp MR. En-gendering choice: preferences for exercising in gender-segregated and gender-integrated groups and consideration of overweight status. Int J Behav Med. 2011 Sep;18(3):216-20. doi: 10.1007/s12529-010-9125-6. PMID 20972657
- [Background] Shapcott KM, Carron AV, Burke SM, Bradshaw MH, Estabrooks PA.Member diversity and cohesion and performance in walking groups. Small Group Research 37, 701-730, 2006.
- [Background] Dunlop WL, Beauchamp MR. Does similarity make a difference? Predicting cohesion and attendance behaviors within exercise group settings. Group Dynamics: Theory, Research, and Practice 15(3): 258-66, 2011.
- [Derived] Beauchamp MR, Liu Y, Dunlop WL, Ruissen GR, Schmader T, Harden SM, Wolf SA, Puterman E, Sheel AW, Rhodes RE. Psychological mediators of exercise adherence among older adults in a group-based randomized trial. Health Psychol. 2021 Mar;40(3):166-177. doi: 10.1037/hea0001060. PMID 33630638
- [Derived] Beauchamp MR, Ruissen GR, Dunlop WL, Estabrooks PA, Harden SM, Wolf SA, Liu Y, Schmader T, Puterman E, Sheel AW, Rhodes RE. Group-based physical activity for older adults (GOAL) randomized controlled trial: Exercise adherence outcomes. Health Psychol. 2018 May;37(5):451-461. doi: 10.1037/hea0000615. PMID 29698019
- [Derived] Beauchamp MR, Harden SM, Wolf SA, Rhodes RE, Liu Y, Dunlop WL, Schmader T, Sheel AW, Zumbo BD, Estabrooks PA. GrOup based physical Activity for oLder adults (GOAL) randomized controlled trial: study protocol. BMC Public Health. 2015 Jun 27;15:592. doi: 10.1186/s12889-015-1909-9. PMID 26116237